CLINICAL TRIAL: NCT00225485
Title: Phase III Study of Effexor XR for the Treatment of Elderly Patients With Depression
Brief Title: Study Evaluating Effexor XR in Elderly Patients With Major Depression.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 0600B1-817
Record Dates: First submitted 2005-09-12; First posted 2005-09-23 (Estimated); Last update posted 2007-05-28 (Estimated); Status verified 2007-05

CONDITIONS: Depression
Keywords: Depression
MeSH Terms: conditions — Depression | interventions — Venlafaxine Hydrochloride

INTERVENTIONS:
Drug: Effexor XR

SUMMARY:
Phase III study evaluating Effexor XR in elderly patients with major depression.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with major depression based on DSM-IV-TR
* Patients having minimal total score of 18 on the HAM-D17 and minimal score of 2 on the item of "depressed mood" of HAM-D at baseline

Exclusion Criteria:

* Patients with schizophrenia or any other psychotic disorder
* Patients with history or presence of bipolar disorder

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 100
Dates: Start 2003-12

PRIMARY OUTCOMES:
Response rate of HAM-D17 (Hamilton Rating Scale for Depression) at the final-on-therapy

SECONDARY OUTCOMES:
Difference of total score of HAM-D17 between baseline and final-on-therapy
Remission rate of HAM-D17 at the final-on-therapy

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (25):
- Japan (25):
  - Ichikawa, Chiba
  - Kasuga, Fukuoka
  - Kitakyushu, Fukuoka
  - Ohnojo, Fukuoka
  - Hiroshima, Hiroshima
  - Otaru, Hokkaido
  - Sapporo, Hokkaido
  - Tsukuba, Ibaragi
  - Hanamaki, Iwate
  - Kawasaki, Kanagawa
  - Sagamihara, Kanagawa
  - Yokohama, Kanagawa
  - Okayama, Okayama-ken
  - Moriguchi, Osaka
  - Sakai, Osaka
  - Sayama, Osaka
  - Adachi-ku, Tokyo
  - Chiyoda-ku, Tokyo
  - Fuchū, Tokyo
  - Higashimurayama, Tokyo
  - Kodaira, Tokyo
  - Meguro-ku, Tokyo
  - Nakano-ku, Tokyo
  - Setagaya-ku, Tokyo
  - Tachikawa, Tokyo